CLINICAL TRIAL: NCT05196997
Title: Construct Validity and Test-Retest Reliability of The De-Morton Mobility Index Turkish Version in Intensive Care Patients
Brief Title: The De-Morton Mobility Index Turkish Version in Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Other Study IDs: DM111
Record Dates: First submitted 2022-01-09; First posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Critical Care; Function; Mobility
Keywords: critical care; function; mobility
MeSH Terms: interventions — Range of Motion, Articular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Mobility and Functional Assessments — The first evaluation was made on the day the patient was discharged from the intensive care unit. DEMMI, Bartel Index, Katz Activities of Daily Living Rating Scale and MRC Muscle Strength Test were performed to the patient, respectively.
  De-Morton Mobility assessment for test-retest reliability was performed again on the 1st day of the patient's service.

SUMMARY:
De Morton Mobility Index is recommended for the evaluation of mobility in the evidence-based guidelines, in patients in intensive care units. The aim of our study is to examine the validity and reliability of the Turkish version of the De Morton Mobility Index in patients hospitalized in the respiratory intensive care unit.

DETAILED DESCRIPTION:
De Morton Mobility Index is recommended for the evaluation of mobility in the evidence-based guidelines, in patients in intensive care units. The aim of our study is to examine the validity and reliability of the Turkish version of the De Morton Mobility Index in patients hospitalized in the respiratory intensive care unit.

Patients aged 18 years and over who were discharged from the ICU were included in our study.

We used De-Morton Mobility Index, Bartel Index, Katz Activities of Daily Living Rating Scale and MRC Muscle Strength Test for convergent validity. De-Morton Mobility assessment for test-retest reliability was performed again on the 1st day of the patient's service.

ELIGIBILITY:
Inclusion Criteria:

* staying in intensive care unit for at least 24 hours
* able to cooperate
* being clinically stable for mobility assessment

Exclusion Criteria:

* the presence of neurological disease
* the presence of orthopedic problems such as fractures
* the presence of metastases
* the presence of cardiorespiratory instability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients aged above 18 years who stayed in the intensive care unit for at least 24 hours and were discharged from the ICU were included in our study.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Mobility Assessment | 15 minutes
  De Morton Mobility Index: It consists of a total of 15 mobility items. The total score ranges from 0-100, with 0 indicating poor mobility and 100 indicating high mobility

SECONDARY OUTCOMES:
Functional independence measurement | 5 minutes
  The Barthel index: It includes 10 items: nutrition, bathroom, personal care, dressing, toilet use, mobility on flat surfaces (immobile, wheelchair use, walking with assistance or independently), transfer (transfer from wheelchair to bed and vice versa), climbing stairs, bowel and bladder continence. It is scored between 0-100. 0; fully independent, 100; means fully independent.
Assessment of daily living activities | 5 minutes
  Katz Index: The index includes basic parameters of daily living activities such as bathing, dressing, toilet, transfer, urine and stool control, nutrition. The scoring of the index varies in the range of 0-6. Higher scores indicate higher independence
Muscle Strength | 10 minutes
  Medical Research Council scale: It includes muscle strength test of six muscle groups. Scoring ranges from 0 to 5 in each muscle group. The maximum score is 60, and a score below 48 indicates significant muscle weakness

CONTACTS AND LOCATIONS:
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naz I, Turgut B, Ediboglu O, Kirakli C. Clinimetric properties of the Turkish version of the De-Morton Mobility Index (DEMMI) in intensive care unit survivors - a cross-sectional observational study. Disabil Rehabil. 2023 Nov;45(22):3730-3736. doi: 10.1080/09638288.2022.2134935. Epub 2022 Oct 20. PMID 36263947